CLINICAL TRIAL: NCT04398875
Title: The Adjunctive Effect of Acupuncture for Advanced Cancer Patients in a Collaborative Model of Palliative Care: a Three-arm Pragmatic Randomized Trial
Brief Title: Adjunctive Effect of Acupuncture for Advanced Cancer Patients With Palliative Care: a Three-arm Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 19-822
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Advanced Cancer
Keywords: advanced cancer; palliative care; acupuncture
MeSH Terms: interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects randomly assigned to either ASC group or SSC group will be blinded to their group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASC (Experimental): Traditional manual acupuncture with standard care (ASC) will be provided. Subjects in the ASC group will receive 9 sessions of acupuncture and standard care for 3 weeks. A semi-standardized acupuncture treatment protocol (combined fixed acupoints with additional acupoints by symptom differentiation) will be employed. The fixed acupuncture points including, Guanyuan (CV4), Xuanzhong(GB39), Sanyinjiao (SP6), Yinlingquan (SP9), Zusanli (ST36), Yingtang (EX-HN3), Baihui (GV20), and Qihai (CV6) will be used in every session.
  Interventions: Other: Acupuncture and standard care (ASC)
- SSC (Sham Comparator): Sham acupuncture plus standard care (SSC) will be provided. Subjects in the SSC group will receive 9 sessions of sham acupuncture and standard care for 3 weeks. The Streitberger sham acupuncture will be employed. The selection of acupoints is the same as ASC.
  Interventions: Other: Sham acupuncture and standard care (SSC)
- SC (Placebo Comparator): Standard care alone (SC) will be provided. Subjects in the SC group will standard care for 3 weeks.
  Interventions: Other: Standard care (SC)

INTERVENTIONS:
Other: Acupuncture and standard care (ASC) — A semi-standardized treatment protocol and standard care will be employed.
  Arms: ASC
Other: Sham acupuncture and standard care (SSC) — Validated non-insertion sham acupuncture (Streitberger sham acupuncture) and standard care will be applied.
  Arms: SSC
Other: Standard care (SC) — Standard care will be employed.
  Arms: SC

SUMMARY:
The proposed study aims to evaluate the adjunctive effect of MA with standard care (ASC) for relieving cancer-related symptoms in a collaborative model of palliative care compared to sham MA plus standard care (SSC) or standard care alone (SC).

DETAILED DESCRIPTION:
After being informed about the study plan, potential risk and benefits, all subjects will give written informed consent prior to participation and undergo eligibility screening. Eligible participants will be randomized into three arms, ASC, SSC, and SC, in a 2:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* All cases are subject to pathology and (or) cytology for a diagnosis of malignant tumour (pathological type is not restricted) at stage IIIB or IV;
* Aged 18 years or above;
* Expected survival time longer than 16 weeks;

Exclusion Criteria:

* Disseminated intravascular coagulation or severe thrombocytopenia with a bleeding tendency, i.e., low platelet count < 35000/µL; INR > 1.5; hemoglobin ≤ 90 g/dL; white blood cell count ≤ 4x109/L;
* Uncontrolled active skin infection;
* Needle phobia;
* Inability to read and understand Chinese;
* Not signed written informed consent.
* Receiving surgery during the whole study period;
* Receiving acupuncture treatment in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of the symptom improvments | Change from baseline score at 3 weeks
  The Edmonton Symptom Assessment System (ESAS) is used to rate the intensity of nine common symptoms experienced by cancer patients. Each symptom is scored from 0 to 10. (0 indicats no symptom and 10 indicates the worst symptom)

SECONDARY OUTCOMES:
EORTC QLQ-C15-PAL | weeks 0, 3, 7 and 11
  The European Organization for Research and Treatment of Cancer Quality of Life 15 items Questionnaire for Palliative Care (EORTC QLQ-C15-PAL)
Numeric Rating Scale | weeks 0, 3, 7 and 11
  The Numeric Rating Scale measures the pain intensity, which is scored from 0-100mm. (no pain at 0 mm, the worst pain at 100mm)
Fatigue | weeks 0, 3, 7 and 11
  The Chinese version of Brief Fatigue Inventory (BFI) is a 9-item, 11-point rating scale developed to assess subjective fatigue.
The Hospital Anxiety and Depression Scale | weeks 0, 3, 7 and 11
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 items. Each item is scored from 0-3. Total score ranges between 0 and 21 for either anxiety or depression.
The Insomnia Severity Index | weeks 0, 3, 7 and 11
  The Insomnia Severity Index (ISI) has 7 items. Each item is sored from 0 to 4. Total scale ranges from 0 t0 28.
Symptom improvments | weeks 0, 1, 2, 7 and 11
  The Edmonton Symptom Assessment System (ESAS) consists of 9 common symptoms experienced by cancer patients. Each symptom is scored from 0 to 10. (0 indicats no symptom and 10 indicates the worst symptom)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyong CHEN, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, So TH, Cho WC, Qin Z, Ma CH, Li SG, Yang Z, Jiang F, Wu J, Zhang ZJ, Kong FM, Lao L. The Adjunctive Effect of Acupuncture for Advanced Cancer Patients in a Collaborative Model of Palliative Care: Study Protocol for a 3-Arm Randomized Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211012749. doi: 10.1177/15347354211012749. PMID 33957783